CLINICAL TRIAL: NCT01242124
Title: Randomized Study of Intrathoracic Side-to-side Stapled Esophagogastric Anastomosis Versus Circular-Stapled Technique in Ivor-Lewis Oesophagectomy
Brief Title: Impact of the Techniques for Intrathoracic Esophagogastric Anastomosis on Outcome in Ivor-Lewis Oesophagectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-CIH-ECC-001
Record Dates: First submitted 2010-11-13; First posted 2010-11-16 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2010-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- side-to-side stapled esophagogastric anastomosis arm (Experimental)
  Interventions: Procedure: side-to-side stapled esophagogastric anastomosis
- circular-stapled esophagogastric anastomosis arm (Active Comparator)
  Interventions: Procedure: circular-stapled esophagogastric anastomosis

INTERVENTIONS:
Procedure: side-to-side stapled esophagogastric anastomosis — 20 patients of distal esophageal cancer receive side-to-side stapled esophagogastric anastomosis in Ivor-Lewis oesophagectomy
  Arms: side-to-side stapled esophagogastric anastomosis arm
Procedure: circular-stapled esophagogastric anastomosis — 20 patients of distal esophageal cancer receive circular-stapled esophagogastric anastomosis in Ivor-Lewis oesophagectomy
  Arms: circular-stapled esophagogastric anastomosis arm

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the side-to-side stapled intrathoracic esophagogastric anastomosis in Ivor-Lewis Oesophagectomy.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the distal esophagus or gastroesophageal junction confirmed by biopsy (squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma) clinical stage I, II, or III.
* Received no previous treatment for esophageal cancer
* Adequate bone marrow, liver and kidney function
* Patients must be able to understand the nature consent of the study and give written informed consent.

Exclusion Criteria:

* Age < 18 years
* History of significant heart disease
* Inoperable on the basis of co-existent medical problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Long and short outcome related with anastomoses | 3 year
  Include anastomotic leakage,anastomotic stricture,regurgitation,heartburn, dumping syndrome and anastomoses diameter.

SECONDARY OUTCOMES:
Quality of life and function outcomes | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: YU zhen tao, M.D., Ph.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin Key Laboratory of Cancer Prevention and Therapy, Tianjin, Tianjin Municipality, China